CLINICAL TRIAL: NCT02254200
Title: Effect of Short-term High-intensity Interval and Fatmax Training on Aerobic and Metabolic Fitness in Obese Subjects
Brief Title: Exercise Training and Fitness in Severe Obesity
Acronym: INTFMOBE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Auxologico Italiano (Other)
Collaborators: University of Lausanne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06C301
Record Dates: First submitted 2014-09-29; First posted 2014-10-01 (Estimated); Last update posted 2015-07-21 (Estimated); Status verified 2015-07

CONDITIONS: Obesity
Keywords: exercise; fat oxidation; indirect calorimetry; insulin sensitivity; weight management
MeSH Terms: conditions — Obesity; Motor Activity; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fatmax group (Experimental): Group who performed a continuous training program at the intensity eliciting the maximal fat oxidation
  Interventions: Other: Fatmax group
- HIIT group (Experimental): Group who performed a continuous training program with high intensity interval
  Interventions: Other: HIIT group

INTERVENTIONS:
Other: Fatmax group — For the Fatmax group each session will consist of 40-50 min of continuous exercise with an intensity that corresponded to the individual Fatmax (moderate intensity)
  Arms: Fatmax group
Other: HIIT group — For HIIT group, each session will consist of 10x60-s cycling intervals interspersed with 60-s of recovery. The workloads will be selected to elicit a heart rate of ~90% maximal heart rate during the intervals with a pedal rate of 90-100 revolutions.min-1, whereas during recovery, the participants will be allowed to pedal against a resistance of 50 W
  Arms: HIIT group

SUMMARY:
Obesity is commonly associated with insulin resistance and hyperinsulinemia, which seem to be linked with an impaired ability to oxidize lipids, particularly in class III obese individuals [Body Mass Index (BMI): > 40 kg*m-2]. Exercise training is an effective strategy to improve insulin sensitivity and to reduce the risk of type 2 diabetes.

This study aimed to compare the effects of two different 2-wk-long training modalities [continuous at the intensity eliciting the maximal fat oxidation (Fatmax) versus adapted high intensity interval training (HIIT)] on aerobic and metabolic fitness of class II and III obese men. It was hypothesized that, because of the nature of HIIT in the stimulation of rapid changes, aerobic fitness, fat oxidation rates during exercise and insulin sensitivity would be improved to a greater extent when adapted HIIT compared to Fatmax training.

DETAILED DESCRIPTION:
Obesity is commonly associated with insulin resistance and hyperinsulinemia, which seem to be linked with an impaired ability to oxidize lipids, particularly in class III obese individuals [Body Mass Index (BMI): > 40 kg*m-2] (1). Exercise training is an effective strategy to improve insulin sensitivity and to reduce the risk of type 2 diabetes (2). It has been suggested that 8 (3) or 10 wk (4) of an individualized moderate exercise training program at intensity (Fatmax) that elicits maximal fat oxidation (MFO) may significantly increase the fat oxidation rates (FORs) during exercise; it may also increase the muscle oxidative capacity in overweight and class I obese men. The effects of an individualized Fatmax training program of a shorter duration have never been investigated.

High-intensity interval training (Wingate-based HIIT) has been shown to induce similar adaptations as traditional training at a moderate intensity following 6 wk of training in healthy adults despite the lower training volume (5). This suggests that HIIT may be a time-efficient alternative (6). Recently, HIIT was also reported to rapidly induce adaptations that are linked to improved health-related outcomes in sedentary and overweight/obese individuals (7, 8).

This study aimed to compare the effects of two different 2-wk-long training modalities [continuous at the intensity eliciting the maximal fat oxidation (Fatmax) versus adapted high intensity interval training (HIIT)] on aerobic and metabolic fitness of class II and III obese men. It was hypothesized that, because of the nature of HIIT in the stimulation of rapid changes, aerobic fitness, fat oxidation rates during exercise and insulin sensitivity would be improved to a greater extent when trained with adapted HIIT compared to Fatmax training.

A group of twenty obese men (BMI≥35 kg*m-2) will be assigned to Fatmax group or to adapted HIIT group. Both groups will perform 8 cycling-sessions matched for mechanical work spread over 14 days [40-50 min continuous exercise at ~60-70% of the maximal heart rate (Fatmax) or 10x60-s cycling intervals a ~90% maximal heart rate interspersed with 60-s recovery (HIIT)]. Aerobic fitness and fat oxidation rates (FORs) during exercise will be assessed prior to and following the training with a maximal incremental test. Blood samples will also be drawn to determine hormones and plasma metabolites levels. Insulin sensitivity was assessed by the homeostasis model assessment of insulin resistance (HOMA).

The experimental design will consist of the following: 1) maximal ramp incremental test, to determine peak power output of each subject. 2) pre training test with blood samples, maximal incremental test (Incr) to determine the whole-body fat oxidation kinetics and Fatmax in the first phase (IncrP1) and the maximal parameters in the second phase (IncrP2) of the test. 3) 2-wk training intervention, Fatmax or HIIT and 4) post-training test, control maximal incremental test with blood samples.

A 3-way repeated-measures ANOVA (time x group x exercise intensity) will be performed to compare the investigated variables.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 35 kg*m-2

Exclusion Criteria:

* Hypertension (blood pressure > 130/90)
* Impaired fasting glucose (> 6.1 mmol*L-1)
* Type 2 diabetes
* Abnormal ECG readings at rest

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2013-01; Primary Completion 2013-12 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Maximal Oxygen consumption (VO2 max) | After two-wk-long of Fatmax or HIIT traning
  VO2 max at incremental test performed at the end of Fatmax or HIIT training period
Fat oxidation rates (FORs) | After two-wk-long of Fatmax or HIIT traning
  FORs at incremental test performed at the end of Fatmax or HIIT training period

SECONDARY OUTCOMES:
HOMA-IR | After two-wk-long of Fatmax or HIIT traning
  Insulin sensitivity assessed by homeostasis model assessment of insulin resistance (HOMA-IR) at the end of Fatmax or HIIT training period
Non-esterified fatty acid (NEFA) | After two-wk-long of Fatmax or HIIT traning
  Resting NEFA at the end of Fatmax or HIIT training period
Insulin | After two-wk-long of Fatmax or HIIT traning
  Resting Insulin at the end of Fatmax or HIIT training period

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Lanzi, MSc, Principal Investigator — University of Lausanne, Department of Physiology; Alberto Salvadori, MD, Study Director — Istituto Auxologico Italiano, Pulmonary Rehabilitation Department; Franco Codecasa, MD, Principal Investigator — Istituto Auxologico Italiano, Pulmonary Rehabilitation Department; Mauro Cornacchia, MD, Study Chair — Istituto Auxologico Italiano, Pulmonary Rehabilitation Department; Davide Malatesta, PhD, Study Director — University of Lausanne, Institute of Sport Sciences; Paolo Fanari, MD, Study Chair — Istituto Auxologico Italiano, Pulmonary Rehabilitation Department
Locations (1):
- Istituto Auxologico Italiano, Ospedale San Giuseppe, Verbania, VB, Italy

REFERENCES:
- [Background] Houmard JA. Intramuscular lipid oxidation and obesity. Am J Physiol Regul Integr Comp Physiol. 2008 Apr;294(4):R1111-6. doi: 10.1152/ajpregu.00396.2007. Epub 2008 Feb 6. PMID 18256136
- [Background] Houmard JA, Tanner CJ, Slentz CA, Duscha BD, McCartney JS, Kraus WE. Effect of the volume and intensity of exercise training on insulin sensitivity. J Appl Physiol (1985). 2004 Jan;96(1):101-6. doi: 10.1152/japplphysiol.00707.2003. Epub 2003 Sep 12. PMID 12972442
- [Background] Dumortier M, Brandou F, Perez-Martin A, Fedou C, Mercier J, Brun JF. Low intensity endurance exercise targeted for lipid oxidation improves body composition and insulin sensitivity in patients with the metabolic syndrome. Diabetes Metab. 2003 Nov;29(5):509-18. doi: 10.1016/s1262-3636(07)70065-4. PMID 14631328
- [Background] Bordenave S, Metz L, Flavier S, Lambert K, Ghanassia E, Dupuy AM, Michel F, Puech-Cathala AM, Raynaud E, Brun JF, Mercier J. Training-induced improvement in lipid oxidation in type 2 diabetes mellitus is related to alterations in muscle mitochondrial activity. Effect of endurance training in type 2 diabetes. Diabetes Metab. 2008 Apr;34(2):162-8. doi: 10.1016/j.diabet.2007.11.006. PMID 18396088
- [Background] Burgomaster KA, Howarth KR, Phillips SM, Rakobowchuk M, Macdonald MJ, McGee SL, Gibala MJ. Similar metabolic adaptations during exercise after low volume sprint interval and traditional endurance training in humans. J Physiol. 2008 Jan 1;586(1):151-60. doi: 10.1113/jphysiol.2007.142109. Epub 2007 Nov 8. PMID 17991697
- [Background] Whyte LJ, Gill JM, Cathcart AJ. Effect of 2 weeks of sprint interval training on health-related outcomes in sedentary overweight/obese men. Metabolism. 2010 Oct;59(10):1421-8. doi: 10.1016/j.metabol.2010.01.002. Epub 2010 Feb 12. PMID 20153487
- [Background] Trilk JL, Singhal A, Bigelman KA, Cureton KJ. Effect of sprint interval training on circulatory function during exercise in sedentary, overweight/obese women. Eur J Appl Physiol. 2011 Aug;111(8):1591-7. doi: 10.1007/s00421-010-1777-z. Epub 2010 Dec 29. PMID 21190036
- [Derived] Lanzi S, Codecasa F, Cornacchia M, Maestrini S, Capodaglio P, Brunani A, Fanari P, Salvadori A, Malatesta D. Short-term HIIT and Fat max training increase aerobic and metabolic fitness in men with class II and III obesity. Obesity (Silver Spring). 2015 Oct;23(10):1987-94. doi: 10.1002/oby.21206. Epub 2015 Sep 3. PMID 26335027